CLINICAL TRIAL: NCT05380674
Title: Health-related Quality of Life in a Cohort of Spanish Schoolchildren and Its Association With the Physical State and Adherence to the Mediterranean Diet.
Brief Title: Health-related Quality of Life in a Cohort of Spanish Schoolchildren.
Status: Completed | Type: Observational
Sponsor: Universidad Católica de Ávila (Other)
Responsible Party: Principal Investigator, JORGE VELAZQUEZ SAORNIL, Principal Investigator, Universidad Católica de Ávila
Other Study IDs: 10/05/2022
Record Dates: First submitted 2022-05-10; First posted 2022-05-19 (Actual); Last update posted 2022-05-19 (Actual); Status verified 2022-05

CONDITIONS: Quality of Life; Physical Inactivity
Keywords: Health-related quality of life; physical state; adherence to the Mediterranean diet; schoolchildren
MeSH Terms: conditions — Sedentary Behavior

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- quality of life: The short questionnaire of healthy habits for adults of the PASOS (Physical Activity, Sedentarism and Obesity in Spanish Youth) study was used, which collects sociodemographic data, weight, height, and physical activity, self-reported.
  Interventions: Behavioral: The short questionnaire of healthy habits

INTERVENTIONS:
Behavioral: The short questionnaire of healthy habits — collects sociodemographic data, weight, height, and physical activity, self-reported.

SUMMARY:
Background: Health-related quality of life (HRQoL) allows knowing the subject's feelings in terms of distress and well-being, as well as her perception of her current and future health.

Objective: Evaluate the associations between health-related quality of life, physical state, and adherence to the Mediterranean diet in a cohort of Spanish children and adolescents. Methods: A cross-sectional study was carried out in a cohort of 305 (47.2% women) children and adolescents aged between 8 and 16 years, in the Primary and Secondary Schools of the province of Ávila (Spain). For the analysis of the different variables, the subjects were classified according to their quality of life in three groups from highest to lowest (Group 1 > Group 2 > Group 3).

ELIGIBILITY:
Inclusion Criteria:

* school children aged 8 to 16
* present the informed consent signed by the parents or legal guardians

Exclusion Criteria:

* serious illness that may influence the nutritional or functional status of the child, mental limitation of the parents and / or children that may hinder the completion of the questionnaire.

Ages: 8 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: school children aged 8 to 16.
Sampling Method: Probability Sample
Enrollment: 305 (Actual)
Dates: Start 2021-01-12 (Actual); Primary Completion 2021-06-01 (Actual); Study Completion 2022-05-01 (Actual)

PRIMARY OUTCOMES:
Health-related quality of life | 3 months
  The descriptive system comprises five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels: no problems, mild problems, moderate problems, severe problems and extreme problems. The patient is asked to indicate their health status by ticking the box next to the most appropriate statement in each of the five dimensions. This decision results in a 1-digit number expressing the level selected for that dimension. The digits of the five dimensions can be combined into a 5-digit number describing the patient's health status.
Eating habits | 3 months
  the total index ranges from 0 to 12, and the final score is classified into three levels:
  >8, ideal Mediterranean diet.
  4-7, improvements needed to adjust the intake to the patterns of the Mediterranean diet.
  ≤3, very poor dietary quality. and adolescence on which the KIDMED index.

CONTACTS AND LOCATIONS:
Locations (1):
- Universidad Católica de Ávila, Ávila, Spain

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Paxton RJ, Jones LW, Rosoff PM, Bonner M, Ater JL, Demark-Wahnefried W. Associations between leisure-time physical activity and health-related quality of life among adolescent and adult survivors of childhood cancers. Psychooncology. 2010 Sep;19(9):997-1003. doi: 10.1002/pon.1654. PMID 19918964
- [Background] Wu XY, Han LH, Zhang JH, Luo S, Hu JW, Sun K. The influence of physical activity, sedentary behavior on health-related quality of life among the general population of children and adolescents: A systematic review. PLoS One. 2017 Nov 9;12(11):e0187668. doi: 10.1371/journal.pone.0187668. eCollection 2017. PMID 29121640
- [Background] Quante M, Kaplan ER, Cailler M, Rueschman M, Wang R, Weng J, Taveras EM, Redline S. Actigraphy-based sleep estimation in adolescents and adults: a comparison with polysomnography using two scoring algorithms. Nat Sci Sleep. 2018 Jan 18;10:13-20. doi: 10.2147/NSS.S151085. eCollection 2018. PMID 29403321
- [Result] Evaristo S, Moreira C, Lopes L, Oliveira A, Abreu S, Agostinis-Sobrinho C, Oliveira-Santos J, Povoas S, Santos R, Mota J. Muscular fitness and cardiorespiratory fitness are associated with health-related quality of life: Results from labmed physical activity study. J Exerc Sci Fit. 2019 Jan 20;17(2):55-61. doi: 10.1016/j.jesf.2019.01.002. Epub 2019 Jan 8. PMID 30740134
- [Result] Muros JJ, Salvador Perez F, Zurita Ortega F, Gamez Sanchez VM, Knox E. The association between healthy lifestyle behaviors and health-related quality of life among adolescents. J Pediatr (Rio J). 2017 Jul-Aug;93(4):406-412. doi: 10.1016/j.jped.2016.10.005. Epub 2017 Jan 25. PMID 28130968
- [Result] Knox E, Muros JJ. Association of lifestyle behaviours with self-esteem through health-related quality of life in Spanish adolescents. Eur J Pediatr. 2017 May;176(5):621-628. doi: 10.1007/s00431-017-2886-z. Epub 2017 Mar 6. PMID 28265762
- [Result] Freedson P, Bowles HR, Troiano R, Haskell W. Assessment of physical activity using wearable monitors: recommendations for monitor calibration and use in the field. Med Sci Sports Exerc. 2012 Jan;44(1 Suppl 1):S1-4. doi: 10.1249/MSS.0b013e3182399b7e. PMID 22157769